CLINICAL TRIAL: NCT03501342
Title: Effects of Immersive Virtual Reality on Balance, Mobility, and Fatigue in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 228
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; virtual reality; balance; mobility; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: prospective randomize controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality group (Experimental): In virtual reality group, 30 minutes of Pilates training, 10 minutes of rest and then 20 minutes of virtual reality will be applied.
  Interventions: Other: Virtual reality group
- Dynamic Balance Training (Active Comparator): In the "Dynamic Balance Training" group, 20 minutes of dynamic balance exercises will be applied after Pilates training.
  Interventions: Other: Dynamic Balance Training
- Control group (No Intervention): The control group will be taught relaxation exercises and will be asked to perform the exercises at home.

INTERVENTIONS:
Other: Virtual reality group — Immersive virtual reality training protocol consisted of "Football" and "Guillotine" games.
  Arms: Virtual reality group
Other: Dynamic Balance Training — Dynamic balance training protocol consisted of holding the ball and running away from the ball with a physiotherapist.
  Arms: Dynamic Balance Training

SUMMARY:
Gait disorder, imbalance, and fatigue are the most frequently reported complaints in Multiple Sclerosis (MS), a chronic neurodegenerative disease. The first symptoms in patients with MS are emerging in the age range 20-50 and these patients need long-term rehabilitation. The virtual reality applications developed for these problems which affect the quality of life negatively and cause disability in the following periods may be a good alternative for conventional rehabilitation applications. In this long-term where motivation is important, virtual reality applications in different environments provide patients with the opportunity to do many different tasks amused. In recent years, the vividness has been increased by the 3D virtual reality headsets.

The aim of this study is to investigate the effects of immersive virtual reality on the balance, mobility, and fatigue in patients with MS.

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized controlled study. The patients will be randomly assigned to three groups, the "immersive virtual reality (IVR)" group, the "dynamic balance training (DBT)" group and the control group. The trainings will be twice a week for 8 weeks. In the IVR group, firstly 30 minutes of Pilates training, 10 minutes of rest and then 20 minutes of virtual reality will be applied. In the DBT group, 20 minutes of dynamic balance exercises will be applied after Pilates training. In dynamic balance training, exercises will consist of similar movements required by virtual reality games. The control group will be taught relaxation exercises and will be asked to perform the exercises 2 times for 8 weeks at home.

Statistical analyses will be performed using the SPSS software version 15 (SPSS Inc. Chicago, IL, USA). The pre-training and post-training measurements of groups will be compared with the Wilcoxon Test. The significance level was set at p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are ambulatory and volunteer to participate to the study, in a stable phase of the disease, without relapses in the last 1 month, with an EDSS between 0-5,5.

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems
* Patients who have any cardiovascular or pulmonary disease in which exercise is contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change between baseline and after 8 weeks of intervention will be assessed
  Berg Balance Scale (BBS) rates performance from 0 (cannot perform) to 4 (normal performance) on 14 items. It has shown to be a valid measure with high inter and interrater reliability for people with MS.

SECONDARY OUTCOMES:
Timed Up and Go Test | Change between baseline and after 8 weeks of intervention will be assessed
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
Modified Sensory Organization Test | Change between baseline and after 8 weeks of intervention will be assessed
  The Modified Sensory Organization Test, which is performed using computerized posturography, measures postural sway in response to 4 different sensory conditions is measured using a force platform.
One-leg standing duration | Change between baseline and after 8 weeks of intervention will be assessed
  One-leg standing duration is measured using chronometer. The time is started when participants lifted a foot from the ground to knee level. The test is terminated when the position disappears or 180 seconds passed.
Activities-specific Balance Confidence | Change between baseline and after 8 weeks of intervention will be assessed
  Activities-specific Balance Confidence (ABC) is a scale in which the patient rates his perceived level of confidence while performing 16 daily living activities.
Fatigue Severity Scale | Change between baseline and after 8 weeks of intervention will be assessed
  In the Fatigue Severity Scale (FSS), participants are asked to rate their fatigue level between 1 and 7 in the 9 statements (including motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life) during the last week.
Fatigue Impact Scale | Change between baseline and after 8 weeks of intervention will be assessed
  Fatigue impact scale consists of forty questions and evaluates the effects of fatigue on the 3 dimensions of daily life activities; cognitive function, physical function and psychosocial function. Each question is graded between 0 (no problem) and 4 (maximum problem).

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Yelnik A, Bonan I. Clinical tools for assessing balance disorders. Neurophysiol Clin. 2008 Dec;38(6):439-45. doi: 10.1016/j.neucli.2008.09.008. Epub 2008 Oct 18. PMID 19026963
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Armutlu K, Keser I, Korkmaz N, Akbiyik DI, Sumbuloglu V, Guney Z, Karabudak R. Psychometric study of Turkish version of Fatigue Impact Scale in multiple sclerosis patients. J Neurol Sci. 2007 Apr 15;255(1-2):64-8. doi: 10.1016/j.jns.2007.01.073. Epub 2007 Mar 6. PMID 17337007